CLINICAL TRIAL: NCT00877799
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Proof of Concept Study to Evaluate the Analgesic Efficacy and Safety of Intravenous CR845 During the Post-Operative Period in Subjects Undergoing Laparoscopic-Assisted Hysterectomy
Brief Title: Study to Evaluate Analgesic Effect of Intravenous Administration of Kappa Agonist CR845 After Hysterectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR845-CLIN2001
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Acute Pain
Keywords: pain; acute pain; visceral pain; kappa agonist; opioid analgesics; peripheral nervous system agents; physiological effects of drugs; surgery; hysterectomy; post-operative; post-operative complications
MeSH Terms: conditions — Acute Pain; Pain; Visceral Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CR845 (Experimental): CR845 administered as a single 15-min i.v. infusion at doses of 0.008 or 0.024 mg/kg on the day after surgery (Cohort 1), or at a dose of 0.040 mg/kg immediately after surgery (Cohort 2)
  Interventions: Drug: CR845
- Placebo (Placebo Comparator): Matched placebo administered as a single 15-min i.v. infusion on the day after surgery (Cohort 1), or the immediately after surgery (Cohort 2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 — CR845 (0.024 mg/kg) administered the day after surgery (Day 1)
  Other Names: Cohort 1: CR845 0.024 mg/kg
  Arms: CR845
Drug: CR845 — CR845 (0.008 mg/kg) administered the day after surgery (Day 1)
  Other Names: Cohort 1: CR845 0.008 mg/kg
  Arms: CR845
Drug: CR845 — CR845 (0.040 mg/kg) administered immediately after surgery (Day 0)
  Other Names: Cohort 2: CR845 0.040 mg/kg
  Arms: CR845
Drug: Placebo — Matched placebo administered the day after surgery (Day 1)
  Other Names: Cohort 1: Matched placebo
  Arms: Placebo
Drug: Placebo — Matched placebo administered immediately after surgery (Day 0)
  Other Names: Cohort 2: Matched placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of single intravenous doses of the kappa opioid agonist CR845 in relieving pain in patients following laparoscopic-assisted hysterectomy surgery. The study protocol was divided into two parts with subjects either dosed with study drug the day following surgery (Cohort 1), or immediately after surgery (Cohort 2).

DETAILED DESCRIPTION:
Currently, the most widely used drugs to treat pain after surgery are opiates, such as morphine. Morphine works mainly by activating one of several types of opiate receptors that control some of our pain sensation - the so-called mu opiate receptors. These receptors are located in many areas of the brain and also outside of the brain. By activating these receptors, morphine provides significant pain relief, but also causes side effects that limit its use. Some of these side effects include: respiratory depression or arrest (slowed or stopped breathing), sedation (a state of calmness or extreme relaxation), euphoria (an exaggerated feeling of physical and mental well-being), constipation, nausea, vomiting, and drug addiction.

In order to avoid the side effects of morphine and other mu opiates, the present experimental drug CR845 was designed to work at a different type of opiate receptor - called kappa - that can also provide pain relief, by acting on sensory nerves outside the brain. CR845 was designed to penetrate the brain much less than other opiate drugs, which should result in pain relief similar to that of morphine, but with fewer side effects. Because CR845 activates kappa receptors instead of mu receptors, the side effects are different than with a morphine-type drug. In particular, kappa opiates, such as CR845, do not cause respiratory depression or arrest, euphoria, constipation, drug tolerance, physical drug dependence or drug addiction. For these reasons, CR845 may present a distinct advantage over other opiates that are currently used for pain relief and post-operative pain in particular.

ELIGIBILITY:
Inclusion Criteria:

* The patients will have an elective laparoscopic-assisted hysterectomy under general anesthesia.
* The patient's preoperative health is graded as the American Society of Anesthesiologists (ASA) risk class of I to III

Exclusion Criteria:

* The patient has a history of known allergies to opioids
* The patient is currently taking opioid analgesics chronically or took opioid analgesics on at least 4 days during the week before surgery.
* Patients having additional procedures (such as those involving the bladder) at the same time as the laparoscopic-assisted hysterectomy.
* Patients taking short-acting oral analgesics (eg, acetaminophen, aspirin, ibuprofen, ketorolac) within 6 hours before administration of study drug; long-acting nonsteroidal anti-inflammatory drugs (NSAIDs) (eg, naproxen, oxaprozin, piroxicam, celecoxib) within 3 days before administration of study drug; systemic steroids within 72 hours before administration of study drug; or any opioid analgesics or tramadol daily for greater than 10 days of the last 30 days before administration of study drug.
* Patients taking the following herbal agents or nutraceuticals within 7 days prior to beginning of the study: chaparral, comfrey, germander, gin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian.
* Patients with clinically significant cardiovascular disease, or cardiac arrhythmias, or significant major risk factors for cardiovascular disease such as poorly controlled hypertension, poorly controlled hypercholesterolemia, poorly controlled diabetes mellitus or serious medical conditions, such as cancer.
* Patient has a history of hepatitis B or C or HIV infection with positive hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibody test.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, Ph.D., Study Director — Cara Therapeutics, Inc.
Locations (12):
- United States (12):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Springhill Medical Center, Mobile, Alabama
  - Helen Keller Hospital, Sheffield, Alabama
  - Paradise Valley Hospital, Phoenix, Arizona
  - Adventist Medical Center, Glendale, California
  - Saddleback Memorial Hospital, Laguna Hills, California
  - Huntington Memorial Hospital, Pasadena, California
  - Palms West Hospital, Loxahatchee Groves, Florida
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - The Ohio State University Medical Center, Columbus, Ohio
  - Memorial Hermann - Memorial City Medical Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two cohorts of patients were enrolled in this study in sequential order. Based on interim analysis of the results for Cohort 1 where study drug was administered 24 hours following surgery, the protocol was revised to administer the study drug immediately following surgery when patients were more likely to report a higher level of pain.
Groups:
- Cohort 1: Placebo: Matched Placebo administered 24 hours post-surgery (Day 1)
- Cohort 1: CR845 0.008 mg/kg: CR845 (0.008 mg/kg) single i.v. dose administered 24 hours post-surgery (Day 1)
- Cohort 1: CR845 0.024 mg/kg: CR845 (0.024 mg/kg) single i.v. dose administered 24 hours post-surgery (Day 1)
- Cohort 2: Placebo: Matched Placebo administered within 3 hours after surgery (Day 0)
- Cohort 2: CR845 0.040 mg/kg: CR845 (0.040 mg/kg) single i.v. dose administered within 3 hours after surgery (Day 0)
Period: Cohort 1: 24 Hours After Surgery (Day 1)
Arm/Group | Cohort 1: Placebo | Cohort 1: CR845 0.008 mg/kg | Cohort 1: CR845 0.024 mg/kg | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Started | 25 | 22 | 21 | 0 | 0
Completed | 22 | 17 | 18 | 0 | 0
Not Completed | 3 | 5 | 3 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 0
Period: Cohort 2: Immediately Post-op (Day 0)
Arm/Group | Cohort 1: Placebo | Cohort 1: CR845 0.008 mg/kg | Cohort 1: CR845 0.024 mg/kg | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Started | 0 | 0 | 0 | 26 | 20
Completed | 0 | 0 | 0 | 24 | 19
Not Completed | 0 | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Placebo: Matched placebo administered within 3 hours post-surgery (Day 0)
- Cohort 2: CR845 0.040 mg/kg: CR845 (0.040 mg/kg) single i.v. dose administered within 3 hours post-surgery (Day 0)
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: CR845 0.008 mg/kg | Cohort 1: CR845 0.024 mg/kg | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg | Total
Number analyzed (Participants) | 25 | 22 | 21 | 26 | 20 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 21 | 26 | 20 | 114
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 21 | 26 | 20 | 114
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 21 | 26 | 20 | 114

OUTCOME MEASURES:

1. Primary Outcome: Responders on Pain Intensity(PI) and Pain Relief (PR) Composite Endpoint
Description: The primary efficacy endpoint was the percentage of treatment responders compared to placebo. A responder was defined as a subject who had at least a 40% reduction in their pain intensity score and a pain relief score of "some," "a lot," or "complete" at 15 and 30 min following the start of the study drug infusion.
Time Frame: 15 and 30 minutes after study drug administration
Population: Results are for Cohort 2 (study drug administered within 3 hours after surgery), ITT population.
Measure: Number; unit: responders
Groups:
- Cohort 2: Placebo: Cohort 2: Matched Placebo administered after surgery on Day 0 when subjects were medically stable and awake with a moderate to severe pain intensity score (i.e., 5 to 8 inclusive on an 11-point NRS) recorded within 3 hr after awakening from anesthesia.
- Cohort 2: CR845 0.040 mg/kg: Cohort 2: CR845 (0.040 mg/kg) administered after surgery on Day 0 when subjects were medically stable and awake with a moderate to severe pain intensity score (i.e., 5 to 8 inclusive on an 11-point NRS) recorded within 3 hr after awakening from anesthesia.
Arm/Group | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Number analyzed (Participants) | 26 | 20
responders | 1 | 1

2. Secondary Outcome: Total PCA Morphine Consumption in the 0-16 Hour Period Following Postoperative Study Drug Treatment
Time Frame: 0 to 16 hours
Population: Results are for Cohort 2 (study drug administered within 3 hours after surgery), ITT population.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Cohort 2: Placebo: Matched Placebo administered within 3 hours after surgery
- Cohort 2: CR845 0.040 mg/kg: CR845 administered within 3 hours after surgery
Arm/Group | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Number analyzed (Participants) | 25 | 20
mg | 24.0 (15.4) | 15.8 (11.8)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: CR845 0.040 mg/kg; Test type: Superiority or Other; p = 0.057, t-test, 2 sided

3. Other Pre Specified Outcome: Total PCA Morphine Consumption in the 4-8 Hour Period Following Postoperative Study Drug Treatment
Time Frame: 4 to 8 hours
Population: Results are for Cohort 2 (study drug administered within 3 hours after surgery), ITT population, based on the number of evaluable patients over the 4-8 hour time interval.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Number analyzed (Participants) | 23 | 19
mg | 5.9 (4.56) | 2.9 (2.63)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: CR845 0.040 mg/kg; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Other Pre Specified Outcome: Total PCA Morphine Consumption in the 8-16 Hour Period Following Postoperative Study Drug Treatment
Time Frame: 8 to 16 hours
Population: Results are for Cohort 2 (study drug administered within 3 hours after surgery), ITT population, based on the number of evaluable patients over the 8-16 hour time interval.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Number analyzed (Participants) | 22 | 19
mg | 6.5 (5.28) | 13.8 (11.5)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: CR845 0.040 mg/kg; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time the patient received her first dose of study drug through the Follow-up Visit.
Groups:
- Cohort 1: Placebo: Matched placebo administered 24 hours after surgery (Day 1)
- Cohort 1: CR845 0.008 mg/kg: CR845 (0.008 mg/kg) administered 24 hours after surgery (Day 1)
- Cohort 1: CR845 0.024 mg/kg: CR845 (0.024 mg/kg) administered 24 hours after surgery (Day 1)
- Cohort 2: CR845 0.040 mg/kg: Cohort 2: CR845 (0.040 mg/kg) administered within 3 hours after surgery (Day 0)
Arm/Group | Cohort 1: Placebo | Cohort 1: CR845 0.008 mg/kg | Cohort 1: CR845 0.024 mg/kg | Cohort 2: Placebo | Cohort 2: CR845 0.040 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/22 | 2/21 | 1/26 | 3/20
Other Adverse Events (participants affected / at risk) | 17/25 | 14/22 | 18/21 | 14/26 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=25) | Cohort 1: CR845 0.008 mg/kg (N=22) | Cohort 1: CR845 0.024 mg/kg (N=21) | Cohort 2: Placebo (N=26) | Cohort 2: CR845 0.040 mg/kg (N=20)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=25) | Cohort 1: CR845 0.008 mg/kg (N=22) | Cohort 1: CR845 0.024 mg/kg (N=21) | Cohort 2: Placebo (N=26) | Cohort 2: CR845 0.040 mg/kg (N=20)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 14 (14) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less